CLINICAL TRIAL: NCT02729181
Title: Assessment of Activities of Daily Living in Adults With Chronic Low Back Pain Using a Nonoperative Treatment Modality: A Retrospective Study
Brief Title: Assessment of Activities of Daily Living in Adults With Chronic Low Back Pain Using a Nonoperative Treatment Modality
Status: Completed | Type: Observational
Sponsor: Integrity Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Axiom-CA-L1N-8R1
Record Dates: First submitted 2016-03-22; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Device: DRX9000

SUMMARY:
The investigators hypothesize that treatment with non-invasive spinal decompression reduces discogenic low back pain (LBP), decreases visual analog pain scale scores, increases activities of daily living and decreases medication use.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* consented to the physician prescribed protocol;
* presented with discogenic low back pain defined as low back pain for minimum of 12 weeks;
* current CT scan

Exclusion Criteria:

* metastatic cancer;
* previous spinal fusion or placement of stabilization hardware within 6 months;
* instrumentation or artificial discs;
* neurologic motor deficits, bladder, or sexual dysfunction;
* alcohol or drug abuse
* patient's with extremes of height (< 147 cm or > 203 cm) and body weight (> 136 kg).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pain Management Clinic
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Lower back pain measured on an 11-point numeric rating scale (VAS) with 0 reflecting no pain at all and 10 the worst imaginable pain. | 12-16 weeks
  0= no pain; 10=worst pain

SECONDARY OUTCOMES:
Functional capacity, measured by activities of daily living | 12-16 weeks
Proportion of patients using adjuvant analgesic medication | 12-16 weeks